CLINICAL TRIAL: NCT04865562
Title: Hormones and Decision Making
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Robert Josephs, Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2015-02-0011
Record Dates: First submitted 2015-02-09; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Dyssocial Behavior
MeSH Terms: conditions — Antisocial Personality Disorder | interventions — Testosterone Propionate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- testosterone (Experimental): 7mg testosterone propionate
  Interventions: Drug: testosterone propionate
- placebo (Placebo Comparator): 125 mg 0.5% cholorbutanol, 50mg saline, pH5
  Interventions: Drug: 0.5% cholorbutanol, saline

INTERVENTIONS:
Drug: testosterone propionate — 1mg/0.1mL solution, to be administered intranasally
  Other Names: Testovis
  Arms: testosterone
Drug: 0.5% cholorbutanol, saline — 125 mg 0.5% cholorbutanol, 50mg saline
  Arms: placebo

SUMMARY:
An investigation of the neuropsychological processes underlying ethical decision making.

DETAILED DESCRIPTION:
This study will investigate the influence of reward sensitivity on cheating behavior via experimental manipulation of reward sensitivity using testosterone.

ELIGIBILITY:
Inclusion Criteria:

* males between 18 and 25

Exclusion Criteria:

* recruitment will be limited to male participants between 18 and 25 years who have no current conditions that would preclude the use of testosterone. Specific exclusion criteria are:
* women of all ages
* males younger than 18 years and older than 25 years
* self-report discomfort with ingestion of testosterone for the purpose of this study
* body mass index lower than 18 or higher than 27
* prior diagnosis of major depression, posttraumatic stress disorder, phobia, anxiety disorder, or other psychiatric conditions
* first-degree relatives diagnosed with a psychiatric disorder
* presence of a medical condition that would preclude the use of testosterone
* use of medications that would preclude the use of testosterone
* consumption of more than 5 cigarettes a day
* current use of testosterone enhancing products, such as gels, creams, and injections

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Measure of ethical behavior - Cheating rate defined as the Average number of 'heads' coin flips participants claim to have obtained | 90 minutes
  drug administration following by behavioral outcome. Specifically, participants will have the opportunity to predict the outcome of a series of coin flips. To obtain a measure of ethical behavior, participants will have the opportunity to cheat by over-reporting their prediction accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Josephs, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- Robert Josephs, Austin, Texas, United States